CLINICAL TRIAL: NCT02769611
Title: A Prospective Phase I/II Dose Escalation Pilot Analysis of Ruboxistaurin (LY333531) for Safety in New York Heart Failure Classification III-IV Patients, As Well As For Efficacy in Acutely Augmenting Cardiac Function.
Brief Title: Ruboxistaurin in New York Heart Failure Classification III-IV Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Tennessee (Other)
Collaborators: The Christ Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-7007
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — ruboxistaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ruboxistaurin 64 mg (Experimental): ruboxistaurin, 64 mg as 1 capsule by mouth with water, 1 time administration
  Interventions: Drug: Ruboxistaurin
- Ruboxistaurin 128 mg (Experimental): ruboxistaurin, 128 mg as 2 capsules by mouth with water, 1 time administration
  Interventions: Drug: Ruboxistaurin
- Ruboxistaurin 256 mg (Experimental): ruboxistaurin, 256 mg as 4 capsules by mouth with water, 1 time administration
  Interventions: Drug: Ruboxistaurin

INTERVENTIONS:
Drug: Ruboxistaurin — Dose escalation trial. 1st ten patients to receive 64 mg, next 10 patients to receive 128 mg, next 10 patients to receive 256 mg.
  Other Names: LY333531

SUMMARY:
This study evaluates the effect of ruboxistaurin for its safety, tolerability, and effectiveness in treating adult patients with heart failure. Patients will receive 1 dose of oral ruboxistaurin.

DETAILED DESCRIPTION:
Ruboxistaurin is a drug initially developed for treatment of diabetic peripheral retinopathy. The proposed indication for ruboxistaurin in this study is the treatment of adult patients with New York Heart Failure Association (NYHA) Class III-IV heart failure. Ruboxistaurin is a protein kinase c-alpha (PKC-alpha) inhibitor and thus will produce an inotropic effect in the heart which holds the potential to improve cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 30-75 years of age, inclusive
2. NYHA Class III-IV heart failure (HF) confirmed left ventricular systolic dysfunction with left ventricular ejection fraction (LVEF) <40% as assessed by noninvasive imaging studies such as echocardiography or cardiac MRI within the last 6 months admitted with decompensated heart failure and almost ready for clinical discharge
3. Patient must have had adequate therapy for acute decompensated HF (heart failure) episode prior to enrollment

Exclusion Criteria:

1. Patients with acute coronary syndrome
2. Resynchronization therapy initiated less than 90 days prior to enrollment
3. (LVAD) left ventricular assist device or heart transplantation expected within the next 3 months
4. Patients on hemodialysis or end stage renal disease (ESRD)
5. Patients with serum albumin less than 3 g/dL or evidence of liver cirrhosis
6. Patients with uncontrolled arterial hypertension (systolic blood pressure > 180 or diastolic blood pressure >110)
7. Patients with severe valvular heart disease
8. Patients with acute myocarditis
9. Patients with serum creatinine >3.0 mg/dl or BUN >70 mg/dL
10. Patients with hemodynamic instability or significant active arrhythmias
11. Patients currently on intravenous inotropic therapy or those that have received inotropic therapy within the last 24 hours prior to study enrollment
12. Patients currently on CYP3A inhibitors, or patients that have taken CYP3A inhibitors within 3 months prior to enrollment
13. Patients with ongoing ischemia
14. Patients who have had a myocardial infarction within 30 days prior to study enrollment
15. Patients who are pregnant, nursing, or planning to become pregnant during the study period

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Percent of patients with a new onset, clinically significant arrhythmia or conduction system disease, | 48 hours
  EKG and continuous holter monitoring will be performed. Determination of clinically significant arrhythmia will be determined by a blinded electrophysiologist; intent to treat population
Percent of patients with significant prolongation in the corrected QT (QTc) interval | 24 hours
  Interpreted by a blinded electrophysiologist. A significant QTc prolongation will be defined as an increase from normal baseline (<440 msec) to greater than 440 msec OR an increase of equal to or more than 5% from baseline for those subjects with a baseline QTc of >440 msec.; Intent to treat population
Percent of patients with significant increase in liver function tests | 12 hours
  An abnormal change in liver function tests will be defined as an increase to 2x the upper limits of normal for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) OR a 50% increase from baseline values. Intent to treat population
Percent of patients with a significant increase in serum creatinine not explained by diuretic use. | 12 hours
  An abnormal change in serum creatinine will be defined as a 50% increase from baseline values. Of note, changes in Blood Urea Nitrogen (BUN) and creatinine may be secondary to diuretic use and intravascular volume depletion. Intent to treat population
Percent of patient with a significant increase in serum creatine phosphokinase (CPK) levels | 12 hours
  An abnormal change in serum CPK will be defined as an increase to 2x the upper limits or normal OR a 50% increase from baseline values. Intent to treat population

SECONDARY OUTCOMES:
Percent of patients experiencing at least one adverse event | 30 days
  Adverse events will be assessed up to 30 days post study drug administration. Intent to treat population
Change in cardiac contractility as assessed by echocardiography. | 4 hours
  Transthoracic echocardiogram performed at baseline and 4 hours. Intent to treat population. Efficacy
Change in self-reported well-being, fatigue and dyspnea | 8 hours, 24 hours
  All subjects will undergo assessment of self-reported global well-being, fatigue and dyspnea via a visual-analogue scale that ranges from 0-100. Intent to treat population

CONTACTS AND LOCATIONS:
Overall Officials: John L Jefferies, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No